CLINICAL TRIAL: NCT01590212
Title: Antenatal Parenting Support for Women Vulnerable in Pregnancy: an Exploratory Randomised Controlled Trial of Mellow Bumps
Brief Title: Mellow Bumps RCT - Antenatal Intervention for Vulnerable Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: Scottish Collaboration for Public Health Research and Policy (Unknown)
Responsible Party: Principal Investigator, Dr Philip Wilson, Professor of Primary Care and Rural Health, University of Aberdeen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12/WS/0024
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Mental Health Wellness 1; Pregnancy; Mother-Child Relations
MeSH Terms: interventions — Pregnancy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Care as usual (No Intervention): Participants received care in line with local guidelines
- Mellow Bumps + care as usual (Active Comparator): MB is a six week group-based antenatal programme designed to support families with additional health and social care needs. MB is intended to decrease maternal antenatal stress levels, increase expectant mothers' understanding of neonates' capacity for social interaction and emphasise the importance of early interaction in enhancing brain development and attachment. It is delivered non-didactically to maximise participant engagement and rapport. Each week there is one activity focused on the woman and another on a baby-related topic. The programme is designed to be offered between twenty to thirty weeks' gestation.
  Interventions: Other: Mellow Bumps
- Chill-out in Pregnancy + care as usual (Active Comparator): CHiP is a relaxation programme that includes all the mother-centred components of Mellow Bumps but none of the baby or mother-baby relationship components. It runs for six weeks at two hours per week. It aims to decrease maternal stress levels.
  Interventions: Other: Chill-out in Pregnancy

INTERVENTIONS:
Other: Mellow Bumps — Mellow Bumps is a six week group-based antenatal programme designed to support families with additional health and social care needs. It is intended to decrease maternal antenatal stress levels, increase expectant mothers' understanding of neonates' capacity for social interaction and emphasise the importance of early interaction in enhancing brain development and attachment. It is delivered non-didactically to maximise participant engagement and rapport. Each week there is one activity focused on the woman and another on a baby-related topic. The programme is designed to be offered between twenty to thirty weeks' gestation, to capture the period when the risk of miscarriage is low and fetal movement felt, but before major preoccupation with the delivery.
  Arms: Mellow Bumps + care as usual
Other: Chill-out in Pregnancy — Chill Out in Pregnancy (ChIP) is a relaxation programme that includes all the mother centred components of Mellow Bumps but none of the baby / mother-baby relationship components. It also runs for six weeks at two hours per week and is intended to decrease stress levels.
  Arms: Chill-out in Pregnancy + care as usual

SUMMARY:
The purpose of this study is to compare the effectiveness of a relationships based antenatal intervention (Mellow Bumps) against a comparison intervention (Chillout In Pregnancy) and also against the normal antenatal care which is received during pregnancy (Care As Usual). The Mellow Bumps intervention will seek to improve maternal anxiety and maternal sensitivity whilst the Chillout In Pregnancy intervention will aim to improve only maternal anxiety. This will allow the researchers to determine what type of intervention, if any, is most successful at improving the outcomes of the mother and child. This will be measured by looking at the mother's stress response, anxiety, depression and irritability, the baby's stress response and the interactions between the mother and the baby. Participants in the study will be pregnant women who would be between 20 and 30 weeks pregnant at the start of the antenatal intervention. Participants will be chosen to take part in one of the three conditions (Mellow Bumps, Chillout In Pregnancy or Care As Usual) at random. All participants will be asked to complete questionnaires and give saliva samples prior to the intervention. The questionnaires will also be repeated at the end of the intervention and at a follow up occurring eight to twelve weeks after birth. Consent will also be sought to take saliva samples from the baby before and after a routine blood test when the baby is five days old. This information will then be evaluated to establish the effectiveness of the proposed interventions.

DETAILED DESCRIPTION:
Lower than anticipated recruitment numbers have resulted in changes to the planned methodology of this trial. Firstly, participants were allocated to the three arms in groups/blocks of 6. Secondly, randomisation of the final group recruited was abandoned.

ELIGIBILITY:
Inclusion Criteria:

* pregnant, between 20 & 30 weeks gestation at start of intervention
* Identified by midwives as meeting Special Needs in Pregnancy (SNiP) criteria
* basic understanding of written and spoken English

Exclusion Criteria:

* not identified as vulnerable through SNiP criteria
* less than 20 weeks or more than 30 weeks gestation at start of intervention

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Wilson, Principal Investigator — University of Glasgow
Locations (2):
- United Kingdom (2):
  - NHS Greater Glasgow & Clyde, Greenock, Inverclyde
  - NHS Ayshire & Arran, Irvine, North Ayrshire

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were identified by community midwifes as having additional health and social care needs in pregnancy in two locations. Recruitment took place between May November 2012.
Pre-assignment Details: Two participants withdrew after randomisation but before baseline data was collected. The researcher was unable to contact two further participants to collect baseline data.
Groups:
- Mellow Bumps + Care as Usual: Mellow Bumps is a targeted intervention aimed at pregnant women with additional health and social care needs.
  Underpinned by attachment theory, there is a focus on:
  Improving maternal wellbeing by reducing stress and anxiety Increasing expectant mother's understandings of neonates' capacity for social interaction Emphasising the importance of early interaction to enhance brain development and attachment.
  Groups meet every week for six weeks when the women is between 20 and 30 weeks pregnant.
- Chill-out in Pregnancy + Care as Usual: Chill-out in Pregnancy is a targeted intervention aimed at pregnant women with additional health and social care needs.
  It is a stress-reduction programme which includes all the mother-centred components of Mellow Bumps but none of the baby or mother-baby relationship elements.
  Groups meet every week for six weeks when the women is between 20 and 30 weeks pregnant.
- Care as Usual: Care-as-usual comprises routine antenatal care provided by the NHS in line with local guidelines.
  Services provided as part of an individividual woman's care plan. If indicated, a pre-birth case conference is held at 28-32 weeks.
Period: Overall Study
Arm/Group | Mellow Bumps + Care as Usual | Chill-out in Pregnancy + Care as Usual | Care as Usual
Started | 12 | 9 | 14
Baseline (Pre-intervention) | 10 (withdrew=2) | 9 | 12 (failed contact=2)
Post-intervention | 7 (failed contact=3) | 6 (failed contact=2; withdrew=1) | 10 (failed contact=1)
Completed | 9 (Includes 2 contacted who failed contact at post-intervention data collection point) | 5 | 9
Not Completed | 3 | 4 | 5
Not completed — Withdrawal by Subject | 2 | 2 | 2
Not completed — Lost to Follow-up | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Two participants withdrew and two were unable to be contacted.
Groups:
- Mellow Bumps (MB) + Care as Usual: MB is a six week group-based antenatal programme designed to support families with additional health and social care needs. MB is intended to decrease maternal antenatal stress levels, increase expectant mothers' understanding of neonates' capacity for social interaction and emphasise the importance of early interaction in enhancing brain development and attachment. It is delivered non-didactically to maximise participant engagement and rapport. Each week there is one activity focused on the woman and another on a baby-related topic. The programme is designed to be offered between twenty to thirty weeks' gestation.
- Chill-out in Pregnancy (CHiP) + Care as Usual: CHiP is a relaxation programme that includes all the mother-centred components of Mellow Bumps but none of the baby or mother-baby relationship components. It runs for six weeks at two hours per week. It aims to decrease maternal stress levels.
- Care as Usual (CAU): Participants received care in line with local guidelines.
- Total: Total of all reporting groups
Arm/Group | Mellow Bumps (MB) + Care as Usual | Chill-out in Pregnancy (CHiP) + Care as Usual | Care as Usual (CAU) | Total
Number analyzed (Participants) | 10 | 9 | 12 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 10 | 8 | 12 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.2 (5.391) | 28.89 (8.594) | 29 (7.851) | 27.14 (7.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 12 | 31
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10 | 9 | 12 | 31
Adult Wellbeing Scale [Mean (Full Range); unit: Scores on a scale] — The Adult Wellbeing scale (AWS): a validated questionnaire which generates scores in four domains - depression, anxiety, outward-directed irritability and inward-directed irritability. The sub-scales have different cut-off scores that indicate a possible problem in that area: Anxiety (normal=0-5, borderline=6-8, problem 9-15), Depression (normal=0-3, borderline=4-6, problem 7-15), Outward directed irritability (normal=0-4, borderline=5-7, problem 8-12), Inward directed irritability (normal=0-3, borderline=4-6, problem 7-12),
  Scores on a scale
    Anxiety | 6.3 [3 to 11] | 6.78 [0 to 12] | 5.36 [0 to 12] | 5.94 [0 to 12]
    Depression | 7.0 [4 to 11] | 6.0 [2 to 10] | 5.0 [1 to 8] | 5.87 [1 to 11]
    Outward directed irritability | 4.8 [1 to 10] | 3.11 [1 to 7] | 3.09 [0 to 6] | 3.65 [0 to 10]
    Inward directed irritability | 2.8 [0 to 6] | 2.33 [0 to 5] | 2.27 [0 to 6] | 2.45 [0 to 6]
Edinburgh Postnatal Depression Scale (EPDS) [Mean (Full Range); unit: Scores on a scale] — Edinburgh Postnatal Depression Scale (EPDS): is a standardised questionnaire which generates a single score. Normal score=0-9, Borderline=10-12, Probable depression=13-30.
  Scores on a scale | 14.10 [8 to 21] | 11 [0 to 20] | 9.27 [1 to 20] | 11.19 [0 to 21]

OUTCOME MEASURES:

1. Primary Outcome: Anxiety, Depression and Irritability Measured on Adult Wellbeing Scale
Description: Anxiety, depression and irritability measured on Adult Wellbeing Scale at 9-12 weeks after baseline.
  The Adult Wellbeing scale (AWS): a validated questionnaire which generates scores in four domains - depression, anxiety, outward-directed irritability and inward-directed irritability. The sub-scales have different cut-off scores that indicate a possible problem in that area: Anxiety (normal=0-5, borderline=6-8, problem 9-15), Depression (normal=0-3, borderline=4-6, problem 7-15), Outward directed irritability (normal=0-4, borderline=5-7, problem 8-12), Inward directed irritability (normal=0-3, borderline=4-6, problem 7-12),
Time Frame: Post intervention (approximately 9-12 weeks after baseline)
Measure: Mean (Full Range); unit: Scores on a scale
Groups:
- Care as Usual: All participants received care in line with local guidelines.
Arm/Group | Mellow Bumps + Care as Usual | Chill-out in Pregnancy + Care as Usual | Care as Usual
Number analyzed (Participants) | 7 | 6 | 10
Scores on a scale
  Depression | 6.57 (3.309) [4 to 13] | 4.67 (2.658) [1 to 8] | 5.50 (2.915) [2 to 10]
  Anxiety | 5.29 (2.563) [3 to 10] | 3.17 (2.714) [0 to 8] | 4.60 (4.061) [0 to 11]
  Outward directed irritability | 3.86 (2.854) [1 to 9] | 2.00 (1.265) [0 to 3] | 2.80 (2.251) [0 to 7]
  Inward directed irritability | 2.14 (1.574) [0 to 4] | 0.83 (0.753) [0 to 2] | 1.20 (1.814) [0 to 6]

2. Primary Outcome: Depression Measured on EPDS
Description: Depression as measured on the EPDS at 9-12 weeks after baseline
  Edinburgh Postnatal Depression Scale (EPDS): is a standardised questionnaire which generates a single score. Normal score=0-9, Borderline=10-12, Probable depression=13-30.
Time Frame: Post-intervention (approximately 9 -12 weeks after baseline)
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Mellow Bumps + Care as Usual | Chill-out in Pregnancy + Care as Usual | Care as Usual
Number analyzed (Participants) | 7 | 6 | 10
scores on a scale | 10.71 (4.957) [7 to 20] | 4.83 (3.251) [1 to 10] | 7.90 (6.887) [0 to 19]

3. Primary Outcome: Anxiety, Depression and Irritability Measured on Adult Wellbeing Scale
Description: Anxiety, depression and irritability measured on the Adult Wellbeing Scale post-birth (approximately 8-12 weeks postnatal)
  The Adult Wellbeing scale (AWS): a validated questionnaire which generates scores in four domains - depression, anxiety, outward-directed irritability and inward-directed irritability. The sub-scales have different cut-off scores that indicate a possible problem in that area: Anxiety (normal=0-5, borderline=6-8, problem 9-15), Depression (normal=0-3, borderline=4-6, problem 7-15), Outward directed irritability (normal=0-4, borderline=5-7, problem 8-12), Inward directed irritability (normal=0-3, borderline=4-6, problem 7-12),
Time Frame: Post-birth (8-12 weeks postnatal)
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Mellow Bumps + Care as Usual | Chill-out in Pregnancy + Care as Usual | Care as Usual
Number analyzed (Participants) | 9 | 5 | 9
scores on a scale
  Depression | 3.44 (1.878) [0 to 6] | 3.44 (2.345) [1 to 7] | 5.14 (4.259) [1 to 10]
  Anxiety | 3.56 (1.944) [0 to 6] | 2.80 (4.087) [0 to 10] | 4.00 (4.822) [0 to 11]
  Outward directed irritability | 2.00 (1.936) [0 to 6] | 1.60 (1.140) [0 to 3] | 2.89 (2.028) [0 to 5]
  Inward directed irritability | 0.89 (1.269) [0 to 3] | 0.80 (1.789) [0 to 4] | 0.67 (1.118) [0 to 3]

4. Primary Outcome: Depression Measured on EPDS
Description: Depression scores as measured on the EPDS post-birth (approximately 8-12 weeks postnatal)
  Edinburgh Postnatal Depression Scale (EPDS): is a standardised questionnaire which generates a single score. Normal score=0-9, Borderline=10-12, Probable depression=13-30.
Time Frame: Post-birth (8-12 weeks postnatal)
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Mellow Bumps + Care as Usual | Chill-out in Pregnancy + Care as Usual | Care as Usual
Number analyzed (Participants) | 9 | 5 | 9
scores on a scale | 5.22 (2.906) [0 to 10] | 2.80 (4.147) [0 to 10] | 5.56 (6.146) [0 to 16]

ADVERSE EVENTS:
Arm/Group | Mellow Bumps + Care as Usual | Chill-out in Pregnancy + Care as Usual | Care as Usual
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/14

LIMITATIONS AND CAVEATS:
Participants lived in one health board area and one community health care partnership (CHCP) in the west of Scotland. Midwives may have approached only those potential participants who were thought to be likely to take part in the group programmes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes